CLINICAL TRIAL: NCT05267873
Title: Combining Data Sources to Identify Effect Moderation for Personalized Mental Health
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Duke University (Other); Patient-Centered Outcomes Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00017538
Record Dates: First submitted 2022-02-20; First posted 2022-03-04 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride; Vortioxetine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Duke Health System Electronic Health Record: Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine
- Johns Hopkins Health System Electronic Health Record: Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine
- Randomized Controlled Trial 1 (NCT01153009): Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine
- Randomized Controlled Trial 2 (NCT01140906): Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine
- Randomized Controlled Trial 3 (NCT00672620): Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine
- Randomized Controlled Trial 4 (NCT00635219): Patients who received Duloxetine or Vortioxetine
  Interventions: Drug: Duloxetine, Vortioxetine

INTERVENTIONS:
Drug: Duloxetine, Vortioxetine — Medications for major depressive disorder

SUMMARY:
This work will extend and apply methods for modeling heterogeneous treatment effects when multiple studies are available, with a particular focus on the complexities in mental health research. The methods will be illustrated in examples estimating the effects of medical treatments for major depressive disorder (duloxetine and vortioxetine) using 4 randomized controlled trials (available in the Vivli trials resource) and non-experimental data from the Duke University Health System electronic health record and the Johns Hopkins Health System electronic health record systems.

ELIGIBILITY:
Duke University Health System Electronic Health Record (EHR) System and Johns Hopkins Health System EHR System

Inclusion criteria:

* All patients prescribed any Duloxetine or Vortioxetine in the health systems between 01/01/2015 - 12/31/2021.
* AND from patients with at least 1-year historical EHR data (burn-in period) without prescribing any of the two medications. During the burn-in period, patients should have at least one encounter in the system, and with no encounters during that time frame when they were prescribed Duloxetine or Vortioxetine.
* AND patients age 18-65 years old at baseline.

Exclusion criteria:

- Patients prescribed both Duloxetine and Vortioxetine at baseline would be removed.

4 randomized controlled trials (RCTs)

Inclusion criteria:

* Male or female
* Age 18 years or older
* Major depressive episode according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) classification code 296.3x
* Montgomery-Asberg Depression Rating Scale (MADRS) total score ≥ 26
* Clinical Global Impression - Severity (CGI-S) scale score ≥ 4

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who received Duloxetine or Vortioxetine
Sampling Method: Non-Probability Sample
Enrollment: 9586 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
9-question Patient Health Questionnaire (PHQ-9) or PHQ-2 scores | 6 months
  Higher score indicates greater severity of major depressive disorder.
9-question Patient Health Questionnaire (PHQ-9) or PHQ-2 scores | 1 year
  Higher score indicates greater severity of major depressive disorder.

SECONDARY OUTCOMES:
Emergency room visits or inpatient admissions with diagnosis of depression or suicidality | 6 months
  A binary outcome equals to 'Yes' if the patient ever had any emergency department or inpatient hospital admission encounter with depression or suicidality International Classification of Diseases (ICD) codes, otherwise equals to "No".
Emergency room visits or inpatient admissions with diagnosis of depression or suicidality | 1 year
  A binary outcome equals to 'Yes' if the patient ever had any emergency department or inpatient hospital admission encounter with depression or suicidality International Classification of Diseases (ICD) codes, otherwise equals to "No".
Emergency room visits or inpatient admissions for any reason | 6 months
  A binary outcome equals to 'Yes' if the patient ever had any emergency department or inpatient hospital admission encounter after the prescription, otherwise equals to "No".
Emergency room visits or inpatient admissions for any reason | 1 year
  A binary outcome equals to 'Yes' if the patient ever had any emergency department or inpatient hospital admission encounter after the prescription, otherwise equals to "No".

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stuart, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Hwanhee Hong, PhD, Principal Investigator — Department of Biostatistics & Bioinformatics, Duke University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No